CLINICAL TRIAL: NCT06224439
Title: Comparison of the Effectiveness of Lumbar Plexus Block and Unilateral Spinal Anaesthesia in Patients Undergoing Femoral Neck Fracture Surgery
Brief Title: Comparison of Regional Anaesthesia Methods for Femoral Neck Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-5/15
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Femoral Neck Fractures; Regional Anesthesia
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hypobaric spinal anaesthesia (Active Comparator): 25 gauge quincke needle will be used for spinal anaesthesia. After the lateral position is given to the patient with the side to be operated on, the patient will be entered through the appropriate interval (L3-4 or L4-5) to apply hypobaric spinal anaesthesia, and after the feeling of falling in the subdural area is obtained, Cerebro Spinal Fluid arrival will be seen and the drug consisting of 0.5% Bupivacain and distilled water with bupivacaine hydrochloride active ingredient will be applied in the range of 2-4cc according to the patient's height and weight.
  Interventions: Procedure: hypobaric spinal anaesthesia
- lumbar plexus block (Active Comparator): A 10-15 cm peripheral block needle, ultrasound and nerve stimulator will be used for lumbar plexus block. Buvicaine with 0.5% Bupivacaine Hydrochloride active substance will be used. It will be diluted half and half with saline. It will be applied in accordance with the patient's height and weight, not exceeding 2mg/kg.
  Interventions: Procedure: lumbar plexus block
- hyperbaric spinal anaesthesia (Active Comparator): 25 gauge quincke needle will be used for spinal anaesthesia. After the lateral position is given to the patient with the side to be operated on, the patient will be entered through the appropriate interval (L3-4 or L4-5) to apply hypobaric spinal anaesthesia, and after the feeling of falling in the subdural area is obtained, Cerebro Spinal Fluid arrival will be seen and the drug consisting of 0.5% hyper Bupivacain hydrochloride active ingredient will be applied in the range of 2-4cc according to the patient's height and weight.
  Interventions: Procedure: hyperbaric spinal anesthesia

INTERVENTIONS:
Procedure: hypobaric spinal anaesthesia — 0.5% Bupivacain and distilled water with bupivacaine hydrochloride active ingredient will be applied in the range of 2-4cc according to the patient's height and weight.
  Arms: hypobaric spinal anaesthesia
Procedure: lumbar plexus block — ultrasound and nerve stimulator will be used for lumbar plexus block
  Arms: lumbar plexus block
Procedure: hyperbaric spinal anesthesia — 0.5% hyperbaric Bupivacain hydrochloride active ingredient will be applied in the range of 2-4cc according to the patient's height and weight.
  Arms: hyperbaric spinal anaesthesia

SUMMARY:
Femoral fracture surgery is frequently performed especially in geriatric population. Compared to general anaesthesia, regional anaesthesia is preferred to general anaesthesia in the geriatric patient population due to lower postoperative pulmonary complications, reduced frequency of delirium and analgesic requirement, intraoperative haemodynamic stability, early postoperative mobilisation and early discharge.

Central and peripheral regional anaesthesia methods have advantages and disadvantages. This situation causes difficulties in the choice of anaesthesia method. Central regional anaesthesia techniques have more haemodynamic effects and higher frequency of complications compared to peripheral methods. The disadvantages of peripheral methods are that they require ultrasound, block needle, nerve stimulator and require knowledgeable and skilled practitioners.

Since there is no study showing the comparison of peripheral nerve blocks and hypobaric spinal anaesthesia with objective nociception values and there are difficulties in the choice of anaesthesia method in this regard, a study was deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* >18 years and <90 years
* ASA (American Society of Anesthesiologists) score between I and IV
* Patients who will undergo femoral neck fracture surgery

Exclusion Criteria:

* Previous local anesthetic allergy
* Those with bleeding diathesis disorder
* Having a mental disorder
* Those who are allergic to the drugs used
* Patients who did not consent to participate in the study
* Presence of infection in the block area
* Body mass index >30
* Preoperative or intraoperative general anesthesia
* Patients for whom consent cannot be obtained
* Pregnant patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-13 (Actual)

PRIMARY OUTCOMES:
intraoperative haemodynamic parameters | intraoperative 2 hours
  non-invasive systolic, diastolic and mean arterial pressure mean arterial pressure (mm/hg)

SECONDARY OUTCOMES:
Entropy | intraoperative 2 hours
  Entropy monitoring involves using electroencephalography-a strip of electrodes applied to the forehead-to assess the depth of general anesthesia in surgical patients. The goal of entropy monitoring is to ensure that patients are given appropriate levels of anesthesia so that recovery is faster. Entropy monitoring provides quantitative measurement of depth of anaesthesia. The Response Entropy scale ranges from 0 (no brain activity) to 100 (fully awake) and the State Entropy scale ranges from 0 (no brain activity) to 91 (fully awake). The clinically relevant target range for entropy values is 40-60.
SPI | intraoperative 2 hours
  The surgical pleth index (SPI) is a dimensionless score which is based on the photoplethysmographic analysis of the pulse wave and the heart beat interval. SPI scores monitored during surgery may reflect a patient's autonomic response to certain nociceptive stimuli. The values of the SPI range from 0 to 100. During general anaesthesia, maintaining a value between 20 and 50 is generally recommended
sedation and analgesic | intraoperative 2 hours
  Intraoperative sedation and analgesic need (Whether there was a need or not how much is given in total mg or mcg)
Intraoperative bleeding | intraoperative 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No